CLINICAL TRIAL: NCT01798147
Title: Selective Internal Radiotherapy (SIRT) Versus Transarterial Chemoembolisation (TACE) for the Treatment of Cholangiocellular Carcinoma (CCC).
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Michael Bernhard Pitton, Consultant, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIRT-TACE-CCC-Mainz-1
Record Dates: First submitted 2013-02-16; First posted 2013-02-25 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Intrahepatic Cholangiocellular Carcinoma
Keywords: Cholangiocellular Carcinoma; TACE; SIRT
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Sirtuins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DEB TACE (Active Comparator): Drug eluting Beads (DC Beads) loaded with Doxorubicin
  Interventions: Procedure: DEB TACE
- SIRT (Experimental): Selective Internal Radiotherapy using Yttrium 90 loaded resin beads (Sir Spheres)
  Interventions: Procedure: SIRT

INTERVENTIONS:
Procedure: DEB TACE — DEB TACE every 6 weeks until either no viable tumor or endpoint reached.
  Other Names: Chemoembolisation
  Arms: DEB TACE
Procedure: SIRT — Selective Internal Radiotherapy once at the beginning of the study. Follow up until endpoint.
  Other Names: Radioembolisation
  Arms: SIRT

SUMMARY:
Selective Internal Radiotherapy is superior to Transarterial Chemoembolisation for the treatment of intrahepatic cholangiocellular carcinoma (CCC).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Intrahepatic CCC, proven by histology or by typical morphology in cross sectional imaging and elevated tumor markers (CEA or CA 19-9)
* Tumor confined to the liver
* At least one measurable lesion in magnetic resonance imaging (MRI)
* Tumor load ≤ 50%
* Preserved liver function (Child Pugh A and B)
* ECOG performance status ≤2

Exclusion Criteria:

* Patients feasible for curative treatment (e.g. resection or local ablation)
* Previous TACE or SIRT
* Prior Chemotherapy
* Child Pugh stage C
* ECOG Performance Status >1
* Tumor involvement >50% of the liver
* Extrahepatic tumor
* Serum Bilirubin >2.0 mg/dl; Serum Albumin 2.8 g/dl, Serum Creatinine >2 mg/dl; Leukocytes <3000/ml; Thrombocytes <50000/ml
* Clinically apparent ascites (ascites only in CT/MRI is no exclusion criteria)
* Esophageal bleeding during the last 3 months
* Hepatic encephalopathy
* Transjugular intrahepatic portosystemic shunt (TIPS)
* Infiltration or occlusion of the main portal vein
* Hepatofugal blood flow in the portal vein
* Hepatopulmonary shunt ≥ 20% in the macroaggregated albumin scan (MAA-scan)
* Contraindications against angiography
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-02; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | at the end of study

SECONDARY OUTCOMES:
Overall survival (OS) | at the end of study
Time to progression (TTP) | at the end of study

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Diagnostic and Interventional Radiology, Mainz, Germany

REFERENCES:
- [Derived] Kloeckner R, Ruckes C, Kronfeld K, Worns MA, Weinmann A, Galle PR, Lang H, Otto G, Eichhorn W, Schreckenberger M, Dueber C, Pitton MB. Selective internal radiotherapy (SIRT) versus transarterial chemoembolization (TACE) for the treatment of intrahepatic cholangiocellular carcinoma (CCC): study protocol for a randomized controlled trial. Trials. 2014 Aug 6;15:311. doi: 10.1186/1745-6215-15-311. PMID 25095718